CLINICAL TRIAL: NCT04763252
Title: Canadian Registry for the Use of Spectrum Therapeutics Cannabis Products in Subjects With Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Canopy Growth Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: #710-4502
Record Dates: First submitted 2021-01-22; First posted 2021-02-21 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Canadian
  Interventions: Other: Spectrum Therapeutics cannabis products

INTERVENTIONS:
Other: Spectrum Therapeutics cannabis products — For the purposes of this study, subjects enrolled will have been authorized Spectrum Therapeutics (ST) products that are commercially available in Canada. The full repertoire of Spectrum Therapeutics products are outlined on the website https://www.spectrumtherapeutics.com/canada/en/patients/products. It encompasses six "colors" (order from Red to Yellow follows the descending THC:CBD ratio), and five types of formulations: soft gels, spray, oil, flowers and vapes). Refer to webpage for the most up to date products available per country https://www.spectrumtherapeutics.com/canada/en/patients/products.

SUMMARY:
Chronic pain affects at least 10% of the global population but is often poorly managed, given the variable efficacy of available pharmacological treatments and the limited accessibility of multidisciplinary interventions. The legalization of cannabis in at least 14 countries and the increasing regulatory approval of cannabis preparations and synthetic cannabinoids and analogues have led to a growing interest in the use of medical cannabis products to manage chronic pain. This use is supported by research demonstrating important interactions between cannabinoids and the human endocannabinoid system and pain modulation pathways. While medical cannabis products are increasingly available to practitioners who treat pain, there is little evidence-based guidance for prescribing or titrating these treatments to manage chronic non-cancer pain. This prospective registry aims to assemble real-world data regarding the use of Spectrum Therapeutics (ST) medical cannabis products in subjects with chronic non-cancer pain in Canada. The registry will also assess treatment outcomes, including pain and related symptoms, global impressions of improvement, and change in concomitant pain medications (opioid use in particular), to better inform the utility of ST products for chronic non-cancer pain management.

Primary Objective:

• To describe patterns of physician selection of Spectrum Therapeutics (ST) medical cannabis treatment regimen, expressed as average daily dose of THC and CBD (in mg), and mode of administration (ingested or inhaled), in the management of chronic non-cancer pain in countries where these products are commercially available.

Secondary Objectives:

* To describe subject product and dose adjustment (under medical follow-up) over time.
* To assess outcomes of treatment, including pain relief and effects on sleep, daily functioning, and quality of life.
* To assess global impressions of treatment effectiveness as reported by subjects and physicians.
* To assess changes in daily dose of opioids, other medications over time.

Safety Objective:

• To assess the safety and tolerability of ST products in subjects with chronic pain.

DETAILED DESCRIPTION:
The present study is a prospective, observational registry designed to generate real-world data on the physician-recommended use of ST products for the management of chronic non-cancer pain in Canada. The study will enroll 500 subjects from 14 sites in geographic regions of ST product distribution, over a 3-year period. Subjects at each site will be followed for one year to collect data on demographics, chronic pain classification, cannabis experience, treatment goals, concomitant medication(s), ST treatment regimen, clinical assessment, subject-reported outcomes, and safety. The study includes five physician-verified visits (baseline, 2, 4, 8, and 12 months), and four at-home subject-verified follow-ups (months 1, 3, 6, 10). Physician verified follow-ups can be conducted in person or via telemedicine. Additionally, should there be a need, according to the physician's judgement, there may be other unscheduled visits, either in-clinic, or via telemedicine. All data will be collected using REDCap Cloud data management platform, via online electronic case report forms (eCRFs), and questionnaires. During physician-verified visits, online questionnaires will be completed by both the physician and the subject (in the presence of a physician or study site personnel). At-home subject-verified follow-ups will be conducted via the REDCap Cloud online portal accessible by computer, tablet, or smartphone.

The following activities will be completed at the Baseline Visit.

* The subject will receive an explanation of the study purpose and procedures, sign the electronic informed consent form (eICF), physician will review eligibility check list, if female of childbearing potential, subject will complete a urine pregnancy test.
* Together, physician and subject will create an account on REDCap Cloud. Together, physician and subject will complete the baseline assessment measuring:

  * Demographics;
  * Chronic pain classification;
  * Cannabis experience;
  * Concomitant medications;
  * Treatment goal;
  * ST treatment regimen;
  * Brief Pain Inventory-Short Form (BPI-SF);
  * Euro Quality of Life Assessment (EQ5D-5L).
* The subject will be scheduled for the first physician-verified follow-up visit approximately 2 months after the initiation of treatment with an ST product.

The following activities will be completed at each physician-verified follow-up visit:

* Physician and subject will discuss the overall treatment regimen.
* Physician will review the subject's online REDCap Cloud entries.
* Together, physician and subject will complete the follow-up visit assessment measuring:

  * ST treatment regimen
  * Concomitant medications
  * Clinician Global Impression of Improvement (CGI-I)
  * BPI-SF
  * EQ5D-5L
  * Patient Global Impression of Change (PGI-C)
  * Physician adverse events (AEs) form

The following measures are to be completed by the subject for each at-home follow-up:

* ST treatment regimen
* Additional cannabis consumption
* BPI-SF
* EQ5D-5L
* Patient Global Impression of Change (PGI-C)
* Subject adverse events (AEs) log

In the event of ST treatment discontinuation or study dropout, physicians will be asked to attempt to follow-up with subjects for the completion of the ST Discontinuation assessment and Exit assessment. Based on physician answers to the ST Discontinuation Assessment, subjects will either stay enrolled in the study (e.g., discontinue all cannabis treatment, but continue to be monitor by site physician for chronic pain), or be withdrawn (e.g., unwilling to stay in the study, switched cannabis licensed producer).

Safety Monitoring:

Spontaneous AE reporting will be entered in REDCap Cloud by the subject during subject follow-ups, using the Subject AE log. Physicians will verify and assess all AEs entered at physician follow-ups, using the Physician AEs form. All serious adverse events will be sent directly to Canopy Growth's Global Pharmacovigilance Department (GPVD) in real-time, where they will be reviewed with respect to country specific regulatory requirements. All non-serious adverse events will be sent in a monthly report to GPVD.

Duration of Subject Participation and Treatment:

Subjects will be followed for one year, unless the subject withdraws early, either independently or in response to physician recommendation. ST treatment will continue for as long as subjects and physicians agree that there is a benefit and treatment is tolerated.

Primary endpoints

* Physician selection of Spectrum Therapeutics (ST) medical cannabis treatment regimen and changes over time in:

  1. average daily dose of THC and CBD (in mg);
  2. route of administration (inhaled or ingested).

     Secondary endpoints
* Subject selection of ST treatment regimen and changes over time in:

  1. average daily dose of THC and CBD (in mg);
  2. route of administration (inhaled or ingested).
* Change in BPI-SF responses from baseline.
* Change in EQ5D-5L responses from baseline.
* PGI-C for the target treatment goal.
* CGI-I for the target treatment goal.
* In subjects taking an opioid, changes in opioid use over time (calculated as milligram morphine equivalents [MME]/day).
* Among subjects taking other medication, total daily dose change over time.

Safety endpoint

• Incidence of AEs stratified by product and formulation.

Number of Subjects (Planned):

Given a continuous enrollment design, the study will include two enrollment milestones over the 3-year study period. Milestone 1, targeted for the end of year 1 (2021) will be to recruit 350 subjects. Milestone 2, targeted for the mid of year 2 (2022) will be to recruit 150 subjects. To enroll a total of up to 500 subjects. The number of subjects may vary based on the real-life use of ST products. Sites will be recruited from countries where ST products are available: Canada, Germany, and Australia. Sites from additional countries may be included as ST products are rolled out in those countries and based on site feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 25 years of age with a diagnosis of chronic non-cancer pain defined as pain lasting or recurring over a period > 3 months (IASP-ICD-11 classification, refer to Appendix 6).
2. Subject is, in the physician's opinion, a candidate for medical cannabis treatment. Candidate status will be determined based on local regulations, common clinical practice, available guidelines and scientific literature, and the physician's expertise or experience with medical cannabis products.
3. Subject received a prescription/authorization for a product in the medical channel of Spectrum Therapeutics.
4. Subject is able to read and understand the informed consent form and complete the study questionnaires.

Exclusion Criteria:

1. Subject refuses to provide informed consent or participate in any aspect of the study.
2. Subject is pregnant or lactating.
3. Subject has a history of psychosis or schizophrenia (or other significant psychiatric disorder), including among first-degree relatives.
4. Subject has a suspected or confirmed cardiovascular disease.
5. Subject is a liver transplant recipient or has severely compromised liver function.

Min Age: 25 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic non-cancer pain patients who received a prescription for a Spectrum Therapeutics medical cannabis product.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Physician selection of Spectrum Therapeutics (ST) medical cannabis treatment regimen and changes over time | Collected at each physician-verified visit (5) over the course of 1-year.
  average daily dose of THC and CBD (in mg); by route of administration (inhaled or ingested).

SECONDARY OUTCOMES:
Subject selection of ST treatment regimen and changes over time in | Collected at each subject-verified visit (4) over the course of 1-year.
  average daily dose of THC and CBD (in mg); by route of administration (inhaled or ingested).
To assess outcomes of treatment including pain relief and effects on sleep | Collected at all follow-ups over the course of 1-year
  Change in Brief Pain Inventory Short Form (BPI-SF) responses from baseline. This is a 9-item self-report questionnaire that includes 6 pain items (e.g., location, 24- hour worst pain, 24-hour average pain, pain right now); 2 treatment items; and 1 (7 part) pain interference item. Minimum value 0 (no pain) and Maximum value 10 (Pain as bas as you can imagine)
To assess outcomes of treatment including daily functioning, and quality of life | Collected at all follow-ups over the course of 1-year
  Change in The EuroQuol Five-Level Quality of Life (EQ5D-5L ) responses from baseline. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions and overall health on a scale from 0-100 (where 100 denotes the best, and 0 the worst health).
To assess global impressions of treatment effectiveness as reported by physicians. | Collected at all follow-ups over the course of 1-year.
  The Clinical Global Impressions of Improvement Scale (CGI-I) for the target treatment goal. A simple question rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment"
To assess global impressions of treatment effectiveness as reported by subjects | Collected at all follow-ups over the course of 1-year.
  The Patient Global Impression of Change scale (PGI-C) for the target treatment goal. A simple question rated on a seven point scale: "Since the start of the study, my overall status is: very much improved; 2=much improved; 3=minimally improved; 4=no change ; 5=minimally worse; 6= much worse; 7=very much worse.
In subjects taking an opioid, changes in opioid use over time | Collected at all physician-verified follow ups over the course of 1-year.
  Calculated as milligram morphine equivalents [MME]/day.
Among subjects taking other medications, changes in use over time | Collected at all physician-verified follow ups over the course of 1-year.
  Calculated as the per day unit specified for the specific medication

OTHER OUTCOMES:
To assess the safety and tolerability of individual ST products in subjects with chronic pain. | Collected at all follow-ups over the course of 1-year
  Incidence of AEs stratified by product and formulation.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Moulin, MD, Principal Investigator — Earl Russell Chair Pain Medicine, Western University
Locations (1):
- Burrard Pain Doctors, Vancouver, British Columbia, Canada

DOCUMENTS (1):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04763252/Prot_000.pdf